CLINICAL TRIAL: NCT03004963
Title: Bioimpedance-guided Fluid Management in Chronic Peritoneal Dialysis Patients: A Randomized Controlled Trial
Brief Title: Bioimpedance-guided Fluid Management in Chronic Peritoneal Dialysis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2016]101K
Record Dates: First submitted 2016-12-12; First posted 2016-12-29 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: End Stage Renal Disease
Keywords: Peritoneal Dialysis; Volume Status; Body Composition Monitor
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- clinical group (Active Comparator): evaluate the volume status just according to clinical indexes in this group.
  Interventions: Device: clinical indexes
- clinical and BCM group (Experimental): Both body composition monitor (BCM) and clinical indexes are used to evaluate the volume status of patients in this group.
  Interventions: Device: Body composition monitor; Device: clinical indexes

INTERVENTIONS:
Device: Body composition monitor — Both body composition monitor (BCM) is used to evaluate the volume status of patients.
  Arms: clinical and BCM group
Device: clinical indexes — The investigators evaluate the volume status of patients according to clinical indexes.

SUMMARY:
Peritoneal dialysis (PD) is one of established treatments in the end stage renal disease patients. Volume overload is a predictor of mortality in PD patients. In this Randomized controlled trial, the investigators use the Body Composition Monitor (BCM), a multifrequency bioimpedance device, to measure the level of overhydration in PD patients and explore its value in fluid management in peritoneal dialysis patients as well as their prognosis.

DETAILED DESCRIPTION:
Optimal fluid management is one of the primary objectives of dialysis treatment, and there is significant concern that peritoneal dialysis (PD) patients can become progressively fluid-loaded with time on treatment, especially as residual kidney function declines. Body Composition Monitor (BCM) has the potential to enable better management of fluid balance. The investigators undertake a prospective, randomized, open-label, controlled trial to determine whether availability of longitudinal BCM measures help clinicians maintain stable fluid status over 24 months in 300 peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older but no older than 80 years.
* who had been on chronic peritoneal dialysis for more than 3 months.
* All of them have signed the informed consent.

Exclusion Criteria:

* were expected to stop PD treatment in 6 months;
* were amputees;
* had a cardiac pacemaker or metallic implants;
* had peritonitis one month before recruitment;
* treated together with hemodialysis;
* were during pregnancy or lactation;
* were positive with HIV;
* had serious diseases, including cancer, infection and liver cirrhosis, which were not suitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
volume status | 96 weeks
  change in overhydration(OH) value
The incidence of cardiovascular events | 96 weeks
  different incidence of cardiovascular diseases
patient mortality | 96 weeks
  different rates of all-cause patient mortality and cardiovascular mortality
technique failure | 96 weeks
  different incidence of technique failure during peritoneal dialysis treatment

SECONDARY OUTCOMES:
blood pressure | 96 weeks
  change in blood pressure
residual renal function | 96 weeks
  decline rate of residual renal function
peritoneal function | 96 weeks
  differences of peritoneal solute transport rate
heart function | 96 weeks
  differences of ejection fraction (EF) in echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Wei Fang, Dr, Principal Investigator — Department of Nephrology, Renji Hospital, Shanghai Jiaotong University, School of Medicine, Shanghai
Locations (1):
- Department of nephrology , Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided